CLINICAL TRIAL: NCT03762343
Title: Ultrasound-guided Greater Occipital Nerve Block in Children Undergoing Posterior Fossa Craniotomy: Randomized, Controlled Study
Brief Title: Ultrasound-guided Greater Occipital Nerve Block in Children Undergoing Posterior Fossa Craniotomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Khaled Abdelfattah Abdallah Sarhan, lecturer of anesthesia, SICU and pain management, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N-11/s /2015/MD
Record Dates: First submitted 2018-11-28; First posted 2018-12-03 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Posterior Fossa Tumor
Keywords: greater occipital nerve block; posterior fossa; ultrasound; pain; craniotomy
MeSH Terms: conditions — Infratentorial Neoplasms; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: An online randomization program (http://www.randomizer.org) will be used to generate random list and to allocate patients into two study groups. Random allocation numbers will be concealed in opaque closed envelops. The patient and investigator performing the block and assessing study outcomes will all be blinded to the study group allocation. The intraoperative study outcomes will be assessed by an anesthetist who is not involved in the block performance and postoperative data will be collected by PICU trained nurses who are blinded to the study groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Greater occipital nerve block group (group GONB) (Experimental): Patient in this group will receive 2 ml of bupivacaine 0.5% (up to a maximum of 2 mg/kg) subcutaneous under ultrasound guidance in the greater occipital nerve region bilaterally.
  Interventions: Drug: ultrasound guided Greater occipital nerve block
- Control group (group C): (Placebo Comparator): Patient in this group will receive the intraoperative standard of care(intraoperative intravenous fentanyl and paracetamol)
  Interventions: Drug: control group C

INTERVENTIONS:
Drug: ultrasound guided Greater occipital nerve block — ultrasound guided Greater occipital nerve block with 2 ml of bupivacaine 0.5% (up to a maximum of 2 mg/kg) subcutaneous under ultrasound guidance in the greater occipital nerve region bilaterally.
  Arms: Greater occipital nerve block group (group GONB)
Drug: control group C — Patient in this group will receive the intraoperative standard of care(intraoperative intravenous fentanyl and paracetamol)
  Arms: Control group (group C):

SUMMARY:
Surgery within the posterior fossa is associated with the highest incidence and greatest severity of acute postoperative pain that may persist beyond the immediate postoperative period.

The utilization of local nerve blocks of the scalp in children may provide analgesia with stable hemodynamics while reducing the need for other anesthetics such as inhaled anesthetics and opioids. This could in turn result in less side effects, higher patient and family satisfaction, and better outcomes.

The use of ultrasound-guided greater occipital nerve block (GONB) for perioperative pain management of posterior fossa surgery in pediatrics is not previously reported.

DETAILED DESCRIPTION:
Surgery within the posterior fossa is associated with the highest incidence and greatest severity of acute postoperative pain that may persist beyond the immediate postoperative period.

Despite a greater awareness of pain after all types of intracranial surgery, clinicians remain reluctant to administer opioids to patients undergoing intracranial surgery because the opioid side effects that may mask signs of neurologic decompensation.

Furthermore, opioids can depress minute ventilation, leading to hypercapnia and increased intracranial pressures. These concerns may be of greater relevance for surgery of the posteriorfossa. However, untreated, pain can also be detrimental. Patients in pain may appear agitated, uncooperative, and experience longer-term pain-related sequelae.

The utilization of local nerve blocks of the scalp in children may thus provide analgesia with stable hemodynamics while reducing the need for other anesthetics such as inhaled anesthetics and opioids: this could in turn result in less side effects, higher patient and family satisfaction, and better outcomes.

The use of ultrasound-guided greater occipital nerve block (GONB) for perioperative pain management of posterior fossa surgery in pediatrics is not previously reported.

The authors hypothesize that ultrasound-guided greater occipital nerve block (GONB) for perioperative pain management of posterior fossa is feasible and superior to conventional methods for perioperative pain management.

After institutional research ethics committee approval, 40 children aged (2-10 years), ASA physical status I or II, Glasgow Coma Scale (GCS) 15, scheduled for craniotomy for posterior fossa tumors will be recruited and a written informed consent will be obtained from the patient guardians.

Anesthetic management:

Patients will not receive any premedication. Upon arrival to the operating room heart rate, noninvasive blood pressure NBP and oxygen saturation SPO2 will be monitored using standard monitor (drȁger infinity vista XL) before inhalational induction of anesthesia using sevoflurane titration (2-8%). 20 or 22 G canula will be inserted after the patient is put to sleep. Anesthesia will be completed by fentanyl (2µg/kg) and atracurium 0.5mg/kg. if IV canula is present anesthesia will be induced by propofol (1-2 mg/kg), fentanyl (2µg/kg) and atracurium 0.5mg/kg After tracheal intubation anesthesia will be maintained using isoflurane 1% in oxygen and air (FIO2 0.6), atracurium infusion at a rate of 0.5 mg/kg/h. Controlled ventilation will be adjusted to maintain moderate hyperventilation (end tidal CO2 30-35 mmHg). A core temperature will be measured using nasopharyngeal probe and a Foley's catheter will be inserted in the urinary bladder. 22G radial arterial canula will be inserted for invasive blood pressure monitoring and blood sampling and central venous line (CVP) will be inserted under complete aseptic condition with ultrasound guidance and wide bore peripheral canula for fluid management.

Greater occipital nerve block:

After the patient is positioned in the prone position with mild neck flexion and after disinfection of the skin; the GON will be located in the short axis plane using the (M-Turbo TM) ultrasound system with a 6-13 MHz high-resolution linear ultrasound transducer (Sonosite, USA).

The ultrasound probe will be placed in a transverse plane over the classical block site, at the level of the superior nuchal line, with the center of the probe at about 2-3 cm lateral to the external occipital protuberance. The GON will be identified in the short axis plane, Then, under real-time scanning, A 22 G canula will be advanced guided with ultrasound using an in-plane (IP) technique from lateral to medial to position the tip of the canula exactly at the center of the nerve. Thereafter, 2 ml of bupivacaine 0.5% will be injected to block the nerve. This technique will then be repeated on the other side.

Vital signs (heart rate, arterial blood pressure, and SpO2) will be monitored continuously And recorded every 30 minutes intraoperatively, and at 2, 4, 6, 8, 12, 16, and 24 hours postoperatively. Bradycardia (heart rate less than 60 beats/minute) will be treated with atropine (0.02mg/kg IV). Fentanyl 0.5 µg /kg as rescue analgesia will be given if HR and systolic BP increased >20% of base line up to maximum 5 µg/ kg. 15 mg/kg of IV paracetamol will be given at the beginning of dural closure at the end of the procedure for both groups.

Postoperative assessment and analgesic regimen:

Objective Pain Scale (OPS) will be assessed at 2, 4, 6, 8, 12, 16, and 24 hours postoperatively. The time to the first request of rescue postoperative analgesic will be: "the time interval between the onset of GONB and the first request to postoperative analgesia and or OPS score ˃2-3". When patients first complain of pain (OPS score ˃2-3) an intravenous paracetamol 15mg/kg will be given and will be repeated every 6 hours. Persistent or breakthrough pain will be managed with incremental intravenous morphine at a dose of 0.05mg/kg to maintain resting OPS at < 2-3. Cumulative 24 hours analgesic consumption will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I or II,
* Glasgow Coma Scale (GCS) 15,
* children scheduled for craniotomy for posterior fossa tumors

Exclusion Criteria:

* Refusal of patients guardians
* Patients with suspected or proved allergic to local anesthetics
* Emergency surgery,
* Children with GCS < 15
* Craniotomy incision beyond the coverage of the block will be excluded from the study.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Objective Pain Scale (OPS) at 12 hours postoperative. | at 12 hours postoperative
  the score has five items(systolic blood pressure, crying, movement,agitation and complain of pain) with a minimum of zero and a maximum of 2 for each item.
  total score = SUM of all points for all parameters
  * Minimum score: 0
  * Maximum score: 10
  * Maximum score if too young to complain of pain: 8 if the score is used with 5 items, a score exceeding the number 3 requires therapeutically effective analgesic. if the score is used with its 4 items, a score exceeding the number 2 requires therapeutic effective analgesic.

SECONDARY OUTCOMES:
Time to first request of postoperative rescue analgesics | within 24 hours
  the time interval between the onset of GONB and the first request to postoperative analgesia and or OPS score ˃2- 3".
Objective Pain Scale (OPS) up to 24 hours. | at 2, 4, 6, 8, 12, 16, and 24 hours postoperatively
  the score has five items(systolic blood pressure, crying, movement,agitation and complain of pain) with a minimum of zero and a maximum of 2 for each item.
  total score = SUM of all points for all parameters
  * Minimum score: 0
  * Maximum score: 10
  * Maximum score if too young to complain of pain: 8 if the score is used with 5 items, a score exceeding the number 3 requires therapeutically effective analgesic. if the score is used with its 4 items, a score exceeding the number 2 requires therapeutic effective analgesic.
Perioperative hemodynamic parameters | every 30 minutes intraoperative and at 2, 4, 6, 8, 12, 16, and 24 hours postoperatively
  Heart rate
side effects | within 24 hours
  number of patients who develop scalp hematoma in the GONB group
side effects | within 24 hours
  number of patients who develop postoperative nausea and vomiting
Perioperative hemodynamic parameters | every 30 minutes intraoperative and at 2, 4, 6, 8, 12, 16, and 24 hours postoperatively
  systolic and diastolic arterial blood pressure.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No